CLINICAL TRIAL: NCT01501734
Title: Bilevel Positive Pressure Ventilation (BIPAP)in Patients With Sleep Disorders Breathing (SDB)and Congestive Heart Failure (CHF):Comparison of Two Diagnostic Methods
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0058-11-MMC
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2012-08

CONDITIONS: Symptomatic Congestive Heart Failure
Keywords: CHF; watch-pat; embletta x; endothelial function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients with symptomatic CHF (Experimental): * Single arm prospective study
  * Study population will include all patients referred to our outpatient clinic for congestive heart failure for a two-year period, who will be screened for sleep apnea and found to have sleep disordering breathing (SDB).
  * 200 patients will visit the outpatient clinic for congestive heart failure.
  * Approximately 30% will be eligible for this study.
  Interventions: Device: watch-pat

INTERVENTIONS:
Device: watch-pat — The Watch-PAT is a home sleep testing (HST) device. The Watch-PAT is a patient-worn, self-contained, non-invasive device used in the patient's home.
  The Watch-PAT diagnoses obstructive sleep apnea (OSA) by measuring the PAT signal, heart rate, oxygen saturation, and actigraphy. The PAT signal is a validated surrogate measure of sympathetic activation that is associated with apneic events and respiratory effort related arousals (RERA). The Watch-PAT provides measures of all the OSA indices, i.e., Apnea Hypopnea Index (AHI), Respiratory Disturbances Index (RDI), and Oxygen Desaturation Index (ODI), which enable accurate assessment of the presence and severity of OSA and its effect on sleep architecture, sleep quality.
  Based on the PAT and actigraphy signals, Watch-PAT differentiates between sleep and wake and detects sleep stages (light, deep, and REM) providing, the effect on additional specific conditions such as REM related apnea.

SUMMARY:
Successful treatment of pulmonary edema was first published in 1938 by A. L. Barach. Since then, this has been the accepted method of treating acute respiratory failure due to left heart failure and edema.

The question was raised if pressure supported ventilation during sleep is used to eliminate sleep apneas, would it be useful also for improving congestive heart failure (CHF). Recent studies assessed the role of continuous positive airway pressure (CPAP) in patients with advanced CHF and found the treatment useful. A possible explanation for these results is that central sleep apnea frequently coexists with severe CHF and is not treated or suppressed by CPAP.

The frequency of central sleep apnea increases with the severity of CHF and can be found in more than 30% of patients.

A few recent studies showed the usefulness of bilevel positive airway pressure (BIPAP) or adaptive servo-ventilation (ASV). ASV led to improvement in ejection fraction as well as in 6 min walking distance testing, and was associated with decreased BNP levels. In another study, bilevel PAP increased LVEF by 7.9%.

The limitations of these studies are the small number of patients and that they were conducted on inpatients only. These factors make it difficult to include BIPAP in the guidelines for chronic heart failure therapy.

Recently, two outpatient modalities have been introduced to diagnose sleep disordering breathing (SDB). However, no study has directly compared the results of both studies in patients with CHF. Moreover, no studies have assessed improvement in CHF after BIPAP treatment.

In addition, the investigators plan to assess the endothelial function in this population before and after BIPAP treatment with the EndoPAT, a noninvasive technology

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients that will be able to sign an informed consent
* Able to use BIPAP equipment
* Established diagnosis of congestive heart failure

Exclusion Criteria:

* Patients who cannot acquire BIPAP from the health care system or who are unable to use the BIPAP.
* Patients who will be not able to visit the clinic for follow up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
changes in frequency of centeral sleep apnea in patients with congestive heart failure before and after BIPAP treatment | 4 months

SECONDARY OUTCOMES:
changes in ejection fraction measured by cardiac echocardiography | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel